CLINICAL TRIAL: NCT03904810
Title: The Effectiveness of Low-frequency High-Intensity Interval Training (HIIT) in Overweight or Obese Young Adults
Brief Title: Low-frequency High-Intensity Interval Training in Overweight or Obese Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIIT001
Record Dates: First submitted 2019-03-31; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Overweight and Obesity
Keywords: HIIT; Exercise frequency; Exercise intensity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: 5 groups ×3 times factorial design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Subjects in this group do not received any intervention
- Moderate Intensity Continuous Training ×3/wk (Active Comparator): Subjects in this group will receive three sessions of Moderate-Intensity Continuous Training per week throughout the 8 weeks experimental period
  Interventions: Behavioral: Exercise intervention
- High Intensity Interval Training×3/wk (Active Comparator): Subjects in this group will receive three sessions of High-Intensity Interval Training per week throughout the 8 weeks experimental period
  Interventions: Behavioral: Exercise intervention
- High Intensity Interval Training×2/wk (Active Comparator): Subjects in this group will receive two session of High-Intensity Interval Training per week throughout the 8 weeks experimental period
  Interventions: Behavioral: Exercise intervention
- High Intensity Interval Training×1/wk (Active Comparator): Subjects in this group will receive one session of High-Intensity Interval Training per week throughout the 8 weeks experimental period
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — HIIT groups performed 30-meter shuttle runs on a rooftop covered field whereas MICT group ran on a footpath with an overall flat and non-slippery road surface. All training sessions were preceded by a 5-minute self-pace warm-up jogging and ended with a 5-minute self-pace jogging or walking cool-down. Each session of MICT consisted of 30 minutes of continuous exercise at an intensity of 60% of heart rate reserve (HRR); [i.e., (maximal HR - resting HR) × intensity + resting HR]. For each HIIT session, the intensity was set at 90% HRR for high-intensity bouts, interspersed with active recovery at 70% HRR. All exercise sessions were supervised by qualified athletic coach or strength and conditioning coach.
  Arms: High Intensity Interval Training×1/wk; High Intensity Interval Training×2/wk; High Intensity Interval Training×3/wk; Moderate Intensity Continuous Training ×3/wk

SUMMARY:
Background: The relationship between the frequency of high-intensity interval training (HIIT) and the resultant adaptations is largely unclear. Purpose: This study examined the effects of different frequencies of HIIT compared to moderate-intensity continuous training (MICT) on body composition and cardiovascular biomarkers in overweight or obese adults. Methods: This study was a randomized, controlled, single-blinded trial. Fifty-six overweight or obese men aged between 18 and 30 years were randomly assigned to no-intervention control (CON; n=14), MICT performed thrice weekly (MICT×3/wk; n=9), HIIT performed thrice weekly (HIIT×3/wk; n=14), HIIT performed twice weekly (HIIT×2/wk; n=10), and HIIT performed once weekly (HIIT×1/wk; n=9). Each HIIT session consisted of 12 × 1-min bouts at 90% heart rate reserve (HRR), interspersed with 11 × 1-min bouts at 70% HRR (HIIT×3/wk: 69 min/wk; HIIT×2/wk: 46 min/wk; HIIT×1/wk: 23 min/wk). Aerobic capacity, resting heart rate, body composition, waist circumference, blood pressure, endothelial function, fasting blood glucose and lipids, circulatory adipokines and inflammatory biomarkers were examined at baseline, after 4 weeks and 8 weeks of intervention.

DETAILED DESCRIPTION:
Individuals who fulfilled the following inclusion criteria were invited to participate in the present study: 1) Chinese male; 2) aged 18-30 years; and 3) overweight or obesity, defined as BMI ≥23 kg/m2 (classification of overweight for Hong Kong adults according to Department of Health, Hong Kong SAR Government) (13). Subjects were excluded if they had: 1) chronic medical and health condition such as cardiovascular diseases, diabetes, neurological disease, musculoskeletal disorder, cancers, and autoimmune diseases; 2) hypertension (blood pressure >140/90 mmHg); 3) contraindications to participating in physical exercise; 4) any pre-existing medical or physical issues that affected the experimental test; 5) physically active (i.e., >3 hours of moderate-intensity exercise weekly) or 6) lean overweight population (BMI ≥23 kg/m2, but percent body fat ≤20%) according to the BMI data corresponding to bioelectrical impedance estimated percent body fat cut-off value among Hong Kong Chinese adults.

Of those who were screened, 103 Chinese young adults were eligible to participate in this study. They were provided with written and verbal information on the study protocol and the possible associated discomforts and risks followed by obtaining their written informed consent to participate in this study. The study protocol and consent form were approved by the Human Subjects Ethics Sub-Committee of The Hong Kong Polytechnic University (ethics approval reference number: HSEARS20160927005-01).

This study was a single-blind, randomized, controlled trial. Subjects were randomly assigned to 1) no-intervention control (CON), 2) MICT performed thrice weekly (MICTx3/wk), 3) HIIT performed thrice weekly (HIITx3/wk), 4) twice weekly (HIITx2/wk), and 5) once weekly (HIITx1/wk). All subjects were instructed to maintain their usual daily activities. Outcome measures including aerobic capacity, body composition, blood pressure, resting heart rate, endothelial function, arterial stiffness, fasting glucose, lipids markers, adipokine marker, and inflammatory marker were assessed at baseline, 4 weeks and 8 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male
2. Aged 18-30 years
3. Overweight or obesity, defined as BMI ≥23 kg/m2 (classification of overweight for Hong Kong adults according to Department of Health, Hong Kong SAR Government)

Exclusion Criteria:

1. Chronic medical and health condition such as cardiovascular diseases, diabetes, neurological disease, musculoskeletal disorder, cancers, and autoimmune diseases
2. Hypertension (blood pressure >140/90 mmHg)
3. Contraindications to participating in physical exercise
4. Any pre-existing medical or physical issues that affected the experimental test
5. Physically active (i.e., >3 hours of moderate-intensity exercise weekly)
6. Lean overweight population (BMI ≥23 kg/m2, but percent body fat ≤20%) according to the BMI data corresponding to bioelectrical impedance estimated percent body fat cut-off value among Hong Kong Chinese adults.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 103 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Estimated maximal oxygen consumption | 8 weeks
  Estimated maximal oxygen consumption achieved during the 20-meter shuttle multistage run test were used for the assessment of aerobic fitness Unit: body weight, estimated oxygen consumption and minute will be combined to report the estimated VO2max in ml/kg/min.
Total running distance | 8 weeks
  Total running distance in meters achieved during the 20-meter shuttle multistage run test were used for the assessment of aerobic fitness
Total body fat percentage | 8 weeks
  Total body fat percentage were assessed by a bioelectrical impedance analyzer (BC-418, Tanita, Japan).
Total body fat mass | 8 weeks
  Total body fat mass in kg were assessed by a bioelectrical impedance analyzer (BC-418, Tanita, Japan).
Total body fat-free mass percentage | 8 weeks
  Total body fat-free mass percentage were assessed by a bioelectrical impedance analyzer (BC-418, Tanita, Japan).
Total fat-free mass | 8 weeks
  Total body fat-free mass were assessed by a bioelectrical impedance analyzer (BC-418, Tanita, Japan).
Trunk fat mass | 8 weeks
  Trunk fat mass in kg were assessed by a bioelectrical impedance analyzer (BC-418, Tanita, Japan).
Body weight | 8 weeks
  Body weight in kg were assessed by a bioelectrical impedance analyzer (BC-418, Tanita, Japan).
Body height | 8 weeks
  Body height in meter were assessed.
Body mass index (BMI) | 8 weeks
  Weight and height will be combined to report BMI in kg/m^2
Waist circumference | 8 weeks
  Waist circumference was determined to the nearest 0.1 cm of a contact tension tape. The tape was applied directly to the skin at the mid-point between the lower margin of the last palpable rib and the top of the iliac crest.

SECONDARY OUTCOMES:
Systolic blood pressure | 8 weeks
  Systolic blood pressure was determined by an electronic sphygmomanometer (Accutorr Plus, Datascope, USA)
Diastolic blood pressure | 8 weeks
  Diastolic blood pressure was determined by an electronic sphygmomanometer (Accutorr Plus, Datascope, USA)
Mean arterial pressure | 8 weeks
  Mean arterial pressure was determined by an electronic sphygmomanometer (Accutorr Plus, Datascope, USA)
Resting heart rate | 8 weeks
  Resting heart rate was determined by an electronic sphygmomanometer (Accutorr Plus, Datascope, USA)
Endothelial function | 8 weeks
  Endothelial function were measured by digital plethysmography using EndoPAT 2000 device (ITAMAR Medical, Caesarea, Israel) and expressed as natural log reactive hyperemia index (LnRHI)
Arterial stiffness | 8 weeks
  Arterial stiffness were measured by digital plethysmography using EndoPAT 2000 device (ITAMAR Medical, Caesarea, Israel) and expressed as augmentation index normalized to heart rate of 75 bpm (AI@75)
Serum fasting glucose | 8 weeks
  Fresh blood samples were sent to an accredited medical laboratory to measure the serum fasting glucose concentrations by commercial test kit methods with an automatic clinical chemistry analyzer (Architect CI8200, Abbott Diagnostics, USA)
Triglycerides | 8 weeks
  Fresh blood samples were sent to an accredited medical laboratory to measure the serum triglycerides concentrations by commercial test kit methods with an automatic clinical chemistry analyzer (Architect CI8200, Abbott Diagnostics, USA)
High-density lipoproteins (HDL) cholesterol | 8 weeks
  Fresh blood samples were sent to an accredited medical laboratory to measure the serum high-density lipoproteins-cholesterol (HDL-C) concentrations by commercial test kit methods with an automatic clinical chemistry analyzer (Architect CI8200, Abbott Diagnostics, USA)
Low-density lipoprotein (LDL) cholesterol | 8 weeks
  Low-density lipoprotein (LDL) cholesterol in serum was measured by an automatic chemistry analyzer (AU-480, Beckman Coulter, USA)
Interleukin 6 | 8 weeks
  Commercially available enzyme-linked immunosorbent assay kits (R&D systems, Minneapolis, MN) were used to determine interleukin 6
Tumor necrosis factor alpha | 8 weeks
  Commercially available enzyme-linked immunosorbent assay kits (R&D systems, Minneapolis, MN) were used to determine tumor necrosis factor alpha
C-reactive protein | 8 weeks
  Commercially available enzyme-linked immunosorbent assay kits (R&D systems, Minneapolis, MN) were used to determine c-reactive protein
Adiponectin | 8 weeks
  Commercially available enzyme-linked immunosorbent assay kits (R&D systems, Minneapolis, MN) were used to determine adiponectin
Intercellular adhesion molecule-1 | 8 weeks
  Commercially available enzyme-linked immunosorbent assay kits (R&D systems, Minneapolis, MN) were used to determine intercellular adhesion molecule-1
Vascular cell adhesion molecule-1 | 8 weeks
  Commercially available enzyme-linked immunosorbent assay kits (R&D systems, Minneapolis, MN) were used to determine vascular cell adhesion molecule-1

CONTACTS AND LOCATIONS:
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No